CLINICAL TRIAL: NCT01653899
Title: Improving Engraftment, Islet Survival and Metabolic Reserve in Clinical Islet Transplantation Using Caspase Inhibitor - IDN-6556
Brief Title: Caspase Inhibition in Islet Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024049
Record Dates: First submitted 2012-07-12; First posted 2012-07-31 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2016-07

CONDITIONS: Diabetes
Keywords: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IDN-6556 (Experimental): Drug
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556 — 14 day oral treatment of the investigational caspase inhibitor drug IDN-6556 following first islet transplant at 50mg twice daily.
  Other Names: Emricasan

SUMMARY:
This is an Investigator Initiated, Phase I/II study, where Type 1 diabetic participants will receive a 14 day oral treatment of the investigational caspase inhibitor drug IDN-6556 following their first islet transplant. Two pilot studies are proposed to establish the optimal safety and efficacy dose of IDN-6556 (25 mg twice daily (Pilot 1) or a loading dose of 100 mg two hours prior to transplantation, then two 50 mg doses following transplant (Day 0) (Pilot 2). This will be followed by 50 mg three times daily). Participants of both pilot studies will receive islet cell transplants under the University of Alberta's standard-of-care therapy.

Secondary objectives include:

1. To determine the proportion of subjects treated with IDN-6556 who achieve and maintain insulin independence after the first or subsequent islet transplant.
2. To obtain preliminary data on the efficacy of IDN-6556 to maintain adequate immunological protection against both allo- and autoimmunity of islet transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

To be eligible the participant must have had T1DM for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

* Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, a Clarke score ≥ 4, HYPO score ≥ 1,000, lability index (LI) ≥ 400 or combined Hypo/LI > 400/300
* Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.

Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

1. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent myocardial infarction (within past 6 months); (b) left ventricular ejection fraction < 30%; or (c) evidence of ischemia on functional cardiac exam.
2. Active alcohol or substance abuse, to include cigarette smoking (must be abstinent for 6 months prior to transplant).
3. Psychiatric disorder making the subject not a suitable candidate for transplantation, (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
4. History of non-adherence to prescribed regimens.
5. Active infection including Hepatitis C, Hepatitis B, HIV, TB (subjects with a positive PPD performed within one year of enrollment, and no history of adequate chemoprophylaxis).
6. Any history of or current malignancies except squamous or basal skin cancer.
7. BMI > 35 kg/m2 at screening visit.
8. Age less than 18 or greater than 68 years.
9. Measured glomerular filtration rate (GFR) < 60 mL/min/1.73 m2.
10. Presence or history of macroalbuminuria (> 300 mg/g creatinine).
11. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
12. Baseline Hb < 105g/L (< 10.5 g/dL) in women, or < 120 g/L (< 12 g/dL) in men.
13. Baseline screening liver function tests outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial LFT panel with any values > 1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
14. Untreated proliferative retinopathy.
15. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast feeding.
16. Previous transplant or evidence of significant sensitization on PRA (at the discretion of the investigator).
17. Insulin requirement > 1.0 U/kg/day
18. HbA1C > 12%.
19. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L (133 mg/dL), treated or untreated; and/or fasting triglycerides > 2.3 mmol/L (90 mg/dL)].
20. Under treatment for a medical condition requiring chronic use of steroids.
21. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5.
22. Untreated Celiac disease.
23. Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the IDN-6556 caspase inhibitor in adult Type 1 diabetic participants receiving their first islet transplant | 3 years post-initial transplant
  The primary objective of this protocol is to assess the safety of the IDN-6556 caspase inhibitor in adult Type 1 diabetic participants receiving their first islet transplant. A tracking log will document adverse events and unexpected complications associated with IDN-6556 using a grading classification as per protocol.

SECONDARY OUTCOMES:
1. To determine the proportion of subjects treated with IDN-6556 who achieve and maintain insulin independence after the first or subsequent islet transplant. | 3 years post-initial transplant
  The proportion of study participants achieving and maintaining insulin independence (c-peptide, HbA1c level) with good glycemic control (blood sugar measurement) at Day 90 and 1, 2, 3 years post-initial islet transplant.
2. To obtain preliminary data on the efficacy of IDN-6556 to maintain adequate immunological protection against both allo- and autoimmunity of islet transplant recipients. | 3 years post-initial transplant
  Immune monitoring for HLA and panel reactive antibody will be performed using serum samples

CONTACTS AND LOCATIONS:
Overall Officials: A.M. James Shapiro, MD PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada